CLINICAL TRIAL: NCT01767519
Title: A Study Evaluating the Efficacy and Safety of BOTOX® or Solifenacin in Patients With Overactive Bladder and Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-125
Record Dates: First submitted 2013-01-11; First posted 2013-01-14 (Estimated); Results first posted 2016-01-12 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Overactive Bladder; Urinary Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Botulinum Toxins, Type A; Solifenacin Succinate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- BOTOX® (Experimental): Treatment Cycle 1: BOTOX injected at Day 1 with one solifenacin placebo capsule taken orally once daily for up to 24 weeks. After a minimum of 12 weeks, patients could request/qualify for a second BOTOX injection.
  Interventions: Biological: BOTOX®; Drug: solifenacin placebo
- solifenacin (Active Comparator): Treatment Cycle 1: Oral solifenacin taken once daily starting at Day 1 for up to 24 weeks with intradetrusor injection of BOTOX placebo on Day 1. After a minimum of 12 weeks, patients could request/qualify for a BOTOX injection.
  Interventions: Biological: BOTOX®; Drug: solifenacin; Drug: Botox placebo (normal saline)
- placebo (Placebo Comparator): Treatment Cycle 1: One solifenacin placebo capsule taken orally once daily starting at Day 1 for up to 24 weeks with an intradetrusor injection of BOTOX placebo at Day 1. After a minimum of 12 weeks, patients could request/qualify for a BOTOX injection.
  Interventions: Biological: BOTOX®; Drug: Botox placebo (normal saline); Drug: solifenacin placebo

INTERVENTIONS:
Biological: BOTOX® — BOTOX 100U injected at Day 1 (BOTOX/solifenacin placebo arm). After a minimum of 12 weeks, all patients could request/qualify for a BOTOX injection.
  Other Names: onabotulinumtoxinA; botulinum toxin Type A
Drug: solifenacin — Beginning on Day 1, one 5 mg solifenicin capsule, with optional dose increase to 10 mg at Week 6, (both overencapsulated for blinding purposes) taken orally once daily for up to 24 weeks.
  Other Names: Vesicare
  Arms: solifenacin
Drug: Botox placebo (normal saline) — Botox placebo (normal saline) intradetrusor injection at Day 1.
  Arms: placebo; solifenacin
Drug: solifenacin placebo — Beginning on Day 1, one capsule taken orally once daily for up to 24 weeks.
  Arms: BOTOX®; placebo

SUMMARY:
A study to evaluate the efficacy and safety of BOTOX® or Solifenacin in patients with overactive bladder (OAB) and urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of Overactive Bladder (OAB) (frequency/urgency) with urinary incontinence for at least 6 months
* Inadequate response or limiting side effects with anticholinergics for the treatment of OAB

Exclusion Criteria:

* Overactive Bladder caused by neurological condition
* Patient has predominance of stress incontinence
* Use of anticholinergics or other medications to treat OAB symptoms in the 7 days prior to screening
* Previous use of solifenacin
* History or evidence of pelvic or urological abnormality
* Previous use of any botulinum toxin of any serotype for any urological condition
* Previous use of any botulinum toxin of any serotype for any non-urological condition within 12 weeks of randomization
* Diagnosis of Myasthenia gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2015-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (8):
- Newport Beach, California, United States
- Leuven, Belgium
- Canada (2):
  - Vancouver, British Columbia
  - Toronto, Ontario
- Prague, Czechia
- Berlin, Germany
- Warsaw, Poland
- London, United Kingdom

REFERENCES:
- [Background] Herschorn S, Kohan A, Aliotta P, McCammon K, Sriram R, Abrams S, Lam W, Everaert K. The Efficacy and Safety of OnabotulinumtoxinA or Solifenacin Compared with Placebo in Solifenacin Naive Patients with Refractory Overactive Bladder: Results from a Multicenter, Randomized, Double-Blind Phase 3b Trial. J Urol. 2017 Jul;198(1):167-175. doi: 10.1016/j.juro.2017.01.069. Epub 2017 Feb 1. PMID 28161352
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant Flow is for Treatment cycle 1, which is the double-blind portion of the study and includes the primary timepoint.
Period: Overall Study
Arm/Group | BOTOX® | Solifenacin | Placebo
Started | 145 | 151 | 60
Completed | 131 | 138 | 55
Not Completed | 14 | 13 | 5
Not completed — Other Reasons | 4 | 4 | 2
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Personal Reasons | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 1 | 2
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Adverse Event | 5 | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BOTOX® | Solifenacin | Placebo | Total
Number analyzed (Participants) | 145 | 151 | 60 | 356
Age, Customized [Number; unit: Participants]
  <65 years | 77 | 79 | 34 | 190
  ≥65 years | 68 | 72 | 26 | 166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 134 | 51 | 308
  Male | 22 | 17 | 9 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Study Baseline in Number of Episodes of Urinary Incontinence in Treatment Cycle 1
Description: Urinary incontinence is defined as involuntary loss of urine as recorded in a patient bladder diary in the 3 consecutive days prior to the study visit in Treatment Cycle 1. The number of incontinence episodes are averaged daily during this period. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Study Baseline, Week 12
Population: Intent-to-Treat: includes all patients according to the group to which they are randomized
Measure: Mean (Standard Deviation); unit: Incontinence Episodes
Arm/Group | BOTOX® | Solifenacin | Placebo
Number analyzed (Participants) | 145 | 151 | 60
Incontinence Episodes
  Study Baseline | 4.86 (3.206) | 5.23 (3.333) | 4.38 (2.485)
  Change from Study Baseline at Week 12 | -3.10 (2.799) | -2.66 (3.059) | -0.98 (2.417)

2. Primary Outcome: Percentage of Patients With 100% Reduction in Incontinence Episodes in Treatment Cycle 1
Description: Urinary incontinence is defined as involuntary loss of urine as recorded in a patient bladder diary in the 3 consecutive days prior to the study visit in Treatment Cycle 1. The number of incontinence episodes are averaged daily during this period and compared to baseline to determine 100% reduction in episodes.
Time Frame: Study Baseline, Week 12
Population: Intent-to-Treat: includes all patients according to the group to which they are randomized
Measure: Number; unit: Percentage of Patients
Arm/Group | BOTOX® | Solifenacin | Placebo
Number analyzed (Participants) | 145 | 151 | 60
Percentage of Patients | 33.8 | 24.5 | 11.7

3. Secondary Outcome: Percentage of Patients With a Positive Response on the Single-Item Treatment Benefit Scale During Treatment Cycle 1
Description: A positive treatment response on the Treatment Benefit Scale is a score of either 1 or 2, representing 'greatly improved' or 'improved.'
Time Frame: Week 12
Population: Intent-to-Treat: includes all patients according to the group to which they are randomized
Measure: Number (95% Confidence Interval); unit: Percentage of Patients
Arm/Group | BOTOX® | Solifenacin | Placebo
Number analyzed (Participants) | 145 | 151 | 60
Percentage of Patients | 71.3 [62.9 to 78.7] | 74.0 [66.1 to 80.9] | 44.8 [31.7 to 58.5]

4. Secondary Outcome: Change From Study Baseline in the Number of Micturition Episodes in Treatment Cycle 1
Description: The number of micturition episodes (the number of times a patient urinates into the toilet) in Treatment Cycle 1 was recorded by the patient in a bladder diary during 3 consecutive days in the week prior to the visit. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Study Baseline, Week 12
Population: Intent-to-Treat: includes all patients according to the group to which they are randomized
Measure: Mean (Standard Deviation); unit: Micturition Episodes
Arm/Group | BOTOX® | Solifenacin | Placebo
Number analyzed (Participants) | 145 | 151 | 60
Micturition Episodes
  Study Baseline | 10.74 (2.520) | 10.40 (2.665) | 10.18 (2.491)
  Change from Study Baseline at Wk 12 (N=135,144,57) | -2.40 (2.827) | -2.03 (2.833) | -0.87 (2.413)

5. Secondary Outcome: Change From Study Baseline in the Number of Nocturia Episodes in Treatment Cycle 1
Description: Nocturia episodes are measured over a 3 day diary prior to each visit in Treatment Cycle 1. A nocturia episode is a void (urinating into the toilet) that interrupts one's sleep. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Study Baseline, Week 12
Population: Intent-to-Treat: includes all patients according to the group to which they are randomized
Measure: Mean (Standard Deviation); unit: Nocturia Episodes
Arm/Group | BOTOX® | Solifenacin | Placebo
Number analyzed (Participants) | 145 | 151 | 60
Nocturia Episodes
  Study Baseline | 2.03 (1.159) | 2.04 (1.083) | 1.98 (0.937)
  Change from Study Baseline at Wk 12 (N=135,144,57) | -0.54 (1.195) | -0.49 (1.133) | -0.23 (1.091)

6. Secondary Outcome: Change From Study Baseline in the Role Limitations Domain on the King's Health Questionnaire in Treatment Cycle 1
Description: The King's Health Questionnaire is a disease-specific questionnaire that measures the quality of life of patients with urinary incontinence. The questionnaire consists of 7 domains, including the role limitations domain. Domain scores range from 0 to 100, with a lower score indicating a preferable health status. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Study Baseline, Week 12
Population: Intent-to-Treat: includes all patients according to the group to which they are randomized
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | BOTOX® | Solifenacin | Placebo
Number analyzed (Participants) | 145 | 150 | 59
Scores on a Scale
  Study Baseline | 76.09 (24.281) [61.1 to 77.2] | 72.11 (26.581) [51.5 to 68.0] | 81.36 (20.781) [39.0 to 66.0]
  Change from Study Baseline at Wk 12 (N=135,145,57) | -30.0 (33.259) [52.0 to 69.0] | -23.79 (31.899) [49.5 to 66.1] | -17.25 (29.033) [29.1 to 55.9]

7. Secondary Outcome: Change From Study Baseline in the Social Limitations Domain on the King's Health Questionnaire in Treatment Cycle 1
Description: The King's Health Questionnaire is a disease-specific questionnaire that measures the quality of life of patients with urinary incontinence. The questionnaire consists of 7 domains, including the social limitations domain. Domain scores range from 0 to 100, with a lower score indicating a preferable health status. A negative number change from baseline indicates an improvement and a positive number change from baseline indicates a worsening.
Time Frame: Study Baseline, Week 12
Population: Intent-to-Treat: includes all patients according to the group to which they are randomized
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | BOTOX® | Solifenacin | Placebo
Number analyzed (Participants) | 145 | 150 | 59
Scores on a Scale
  Study Baseline | 59.66 (21.442) [61.1 to 77.2] | 56.22 (22.708) [51.5 to 68.0] | 62.57 (22.551) [39.0 to 66.0]
  Change from Study Baseline at Wk 12 (N=135,145,57) | -13.46 (21.906) [52.0 to 69.0] | -12.70 (21.361) [49.5 to 66.1] | -7.60 (21.667) [29.1 to 55.9]

ADVERSE EVENTS:
Description: The safety population includes all patients who received at least 1 dose of study medication. The safety population is used to assess adverse events and serious adverse events. Adverse events and serious adverse events are displayed for the placebo-controlled treatment Cycle 1.
Arm/Group | BOTOX® | Solifenacin | Placebo
Serious Adverse Events (participants affected / at risk) | 6/145 | 6/147 | 2/60
Other Adverse Events (participants affected / at risk) | 57/145 | 40/147 | 13/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | BOTOX® (N=145) | Solifenacin (N=147) | Placebo (N=60)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Polysubstance dependence (Psychiatric disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/123 | 1/131 | 0/51 — FEMALE ONLY
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BOTOX® (N=145) | Solifenacin (N=147) | Placebo (N=60)
Dry mouth (Gastrointestinal disorders) | 4 | 12 | 0
Urinary tract infection (Infections and infestations) | 37 | 15 | 6
Bacteriuria (Infections and infestations) | 11 | 14 | 3
Residual urine volume (Investigations) | 10 | 0 | 1
Urinary retention (Renal and urinary disorders) | 10 | 1 | 0
Dysuria (Renal and urinary disorders) | 6 | 8 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.